CLINICAL TRIAL: NCT06753058
Title: ERAS Protocol on Maternal and Fetal Outcomes Following Elective Cesarean Section: a Controlled Trial
Brief Title: ERAS Protocol on Maternal and Fetal Outcomes Following Elective Cesarean Section
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Berrin Gunaydin, Professor, MD, PhD, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Decision no: 502/31.05.2021
Record Dates: First submitted 2024-12-05; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pregnant Women; Enhanced Recovery After Surgery (ERAS) Protocol
Keywords: enhanced reocery after surgery; obstetric quality -of-recovery score; cesarean section; spinal anesthesia; newborn well being

STUDY DESIGN:
Intervention Model Description: In this interventional study, Enhanced Recovery After Surgery (ERAS) protocol for cesarean has been planned to apply to the parturients who accepted to participate to the study.
  Unfortunately randomization cannot be done since the strategy for assigning participants to apply ERAS intervention was based on the obstetric team's preference first. The rest of the parturients were regarded as the control group (standard care) who did not receive ERAS intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STANDARD CARE (CONTROL) (No Intervention): Standard care as control includes ROUTINE preoperative, peroperative and postoperative approach of the institution for the management of cesraean delivery under spinal anesthesia.
- ERAS PATHWAY (Experimental): ERAS INTERVENTION includes 3 steps:
  1. preoperative components (face to face education/information about fasting, Cesarean Section and/or anesthesia, antimicrobial prophylaxis, breastfeeding preparation and support, fasting schedule, anemia screening-hemoglobin optimization if needed),
  2. peroperative components (antibiotic and antiemetic prophylaxis, management of neuraxial anesthesia, maintenance of normothermia, uterotonic use), 3. postoperative components (early oral intake/urinary catheter removal/mobilization, early mother-newborn bonding and encouraged breastfeeding).
  Interventions: Dietary Supplement: 25 gram of maltodextrin in 330 mL , Nutricia Fantomalt 4 Gram, Nutri Gıda Ürünleri San. ve Tic. A.Ş., Istanbul, Türkiye, 2 h prior to surgery.; Behavioral: Mother baby bonding

INTERVENTIONS:
Dietary Supplement: 25 gram of maltodextrin in 330 mL , Nutricia Fantomalt 4 Gram, Nutri Gıda Ürünleri San. ve Tic. A.Ş., Istanbul, Türkiye, 2 h prior to surgery. — Although 45 g of different carbohydrate solutions either Gatorade 54 g carbohydrate or clear apple juice 56 g carbohydrate in non-diabetic women have been recommended by SOAP, we preferred 25 g of carbohydrate, fantomalt, nutricia, diluted in the 330 mL in both diabetic and non-diabetic pregnant women.
  Arms: ERAS PATHWAY
Behavioral: Mother baby bonding — In the ERAS implemented group, mother-baby contact to promote early bonding was established, and both mother and baby were encouraged for breastfeeding. In the control group, only mother-baby contact was facilitated without proactive breastfeeding encouragement.
  Arms: ERAS PATHWAY

SUMMARY:
The goal of this observational study is to investigate the maternal, fetal, and neonatal outcomes in parturients scheduled to undergo elective cesarean section (CS) receiving either standard care or enhanced recovery after surgery (ERAS) protocol.

Primary purpose is to learn if implementing ERAS protocol can improve maternal outcomes in pregnant women aged greater than 18 years scheduled to undergo elective CS under spinal anesthesia using patient reported outcome mesaure (PROM).

Secondary purpose is to learn if implementation of maternal ERAS protocol can improve neonatal outcome in terms of nutrition and breastfeeding.

The main questions that aims to answer are maternal recovery outcome measure determined by obstetric quality recovery score (ObsQoR) which has been known as a patient reported outcome mesaure (PROM) and neonatal outcome assessed by pediatricians.

Primary outcome measure is improved maternal recovery in term of ObsQoR in the ERAS pathway.

Secondary outcome measure is improved neonatal outcome in terms of nutrition and breastfeeding in the ERAS pathway.

DETAILED DESCRIPTION:
Methods After obtaining approval of the institutional ethics committee (Decision number: 502/Date: 31.05.2021) and written informed consent from the parturients, data were collected prospectively in 450 ASA II or III term pregnant women aged ≥18 years scheduled to undergo elective CS under spinal anesthesia between June 2021 and June 2023. Gazi University Hospital, which is a re-accredited tertiary care referral center by ESAIC (European Society of Anaesthesiology and Intensive Care), has an annual rate of approximately 1400 deliveries. Parturients younger than <18 years old with fetal compromise, ASA IV or V physical status and emergency cases were not included in this study. The ERAS protocol introduced for our unit was adapted from the SOAP. Following approval of the ERAS protocol by the obstetric team and the participants, two groups were assigned as; ERAS group (n=150) and control group (n=300) who would receive standard care of the unit. The data of the parturients having standard care were compared with those who were enrolled in the ERAS pathway.

Features of ERAS implementation and standard care in the study Step 1. Preoperative (Antepartum) Components

1. Enrolled patients were seen in the antenatal clinic to give face to face education including information about fasting, CS and/or anesthesia, antimicrobial prophylaxis, skin washing, breastfeeding preparation and support by the principal researcher anesthesiologist for ERAS pathway to improve patient understanding and engagement in their own care.
2. Principally fasting 6 hours (h) for solids and 2 h for clear fluids was provided. To standardize fasting duration according to the scheduled time of surgery in the ERAS group, parturients who were scheduled for CS before 12:00 PM were allowed to have breakfast at 2:00 AM, while the rest scheduled for CS after 12:00 PM were allowed to have breakfast at 6:00 AM. On the morning of surgery, parturients either diabetic or non-diabetic in the ERAS implemented group were given a carbohydrate solution prepared by the principal researcher anesthesiologist containing 25 g of maltodextrin in 330 mL approximately 2 h prior to surgery.

   The control group fasted after 12:00 AM regardless of the scheduled CS time and no carbohydrate solution was administered prior to surgery.
3. Anemia screening and treatment for hemoglobin optimization was done in both groups.

Step 2. Perioperative (Intrapartum) Components

1. Standard intravenous (IV) antibiotic prophylaxis as per hospital guidelines was done in both groups (IV Cefazolin 2 gram in case of no known allergy history).
2. Management of anesthesia/analgesia (neuraxial 100 microgram of morphine and 10 microgram of fentanyl), maintenance of fluid and surgical techniques were similar in both groups. As per our obstetric anesthesia division practice [16], weight-height adjusted dose of hyperbaric bupivacaine 0.5% with morphine plus fentanyl was used during co-loading of 500 mL of colloid (VOLUHES, HES 130/0.4, 6% I.V., Polifarma, Türkiye) for spinal anesthesia and spinal anesthesia induced hypotension was treated with 10 mg of ephedrine (only available vasopressor drug in the country) in IV bolus doses in both groups.
3. Despite all parturients in both groups received 10 mg of IV metoclopramide prophylactically, parturients in the ERAS implemented group received IV 1.5 mg of the 5-HT3 antagonist granisetron additionally. In both groups, in case of risk factors for intraoperative and postoperative nausea and vomiting (PONV), IV 4 mg of dexamethasone was added.
4. To maintain normothermia body temperature loss was prevented using under-patient-mattress-blankets and warmers along with the control of the operating theatre temperature.
5. After the delivery of the baby, uterotonics were administered as per hospital guidelines (50 microgram of carbetocin IV bolus was given and followed by 20 IU of oxytocin in 1000 ml of normal saline infusion was started at a rate of 2.5-7.5 IU/ hour) in both groups.

Delayed cord clamping was not performed in any of the groups by the obstetricians.

Step 3. Postoperative Components

1. In both groups who are at risk for deep vein thrombosis, prophylaxis was provided using pneumatic compression stockings.
2. Blood glucose monitoring was conducted only in diabetic patients and those with symptoms of hypoglycemia during follow-up.
3. In the ERAS implemented group, the diet management plan was as follows:

   * drinking clear water was started at 2 h postoperatively
   * eating liquid diet (regime I or II) was started at 4 h

     * Regime I (R-I) is a clear liquid diet that contains pulp-free, grain-free liquid drinks such as sweetened tea, fruit juice, compote water, lemonade, meat and chicken broth.
     * Regime II (R-II) is a soft diet that consists of soft, easily chewable and digestible foods such as; light soups, mashed and boiled potatoes, puddings and liquid drinks, etc.
   * eating normal diet (regime III-IV) was started at 6 h

   In the control group, the oral intake -diet management plan was as follows:
   * drinking water at 6 h postoperatively
   * eating diet R I-II a few h later
   * eating diet R III-IV after 1st flatus
4. Parturients in the ERAS implemented group were encouraged to chew gum with early feeding, while patients in the control group were not.
5. The urinary catheter was removed just before mobilization in the ERAS implemented group, whereas it was removed when urine output reached to 1000 mL as per clinical conventional procedure in the control group.
6. In the ERAS implemented group, mother-baby contact to promote early bonding was established, and both mother and baby were encouraged for breastfeeding. In the control group, only mother-baby contact was facilitated without proactive breastfeeding encouragement.
7. Prior to discharge, both groups were asked to fill out the validated Turkish version of the ObsQoR-11 with 11-point Likert scale. These forms were collected.

Recorded parameters;

* maternal demographics, comorbidities with medications and history (drug allergy, surgical and obstetric)
* preoperative duration of fasting for fluid and solid food, time to intake of 1st postoperative water, regimen I-II and regimen III-IV
* time to mobilization, urinary catheter removal and flatus and LOS for mother (in hours)
* postoperative pain within 24 h of the surgery was assessed for all patients using VAS scores at postoperative 24 h in rest and extra analgesic requirement
* validated Turkish version of 11-item ObsQoR score with an 11-point numerical Likert scale (0 being strongly negative, 10 being strongly positive) resulting maximum score of 110.
* postoperative complications (hypoglycemia, hypotension, PONV)
* newborn demographics and Apgar scores, umbilical cord gas analysis, newborn LOS in days
* need for follow-up in the ward or newborn intensive care unit (NICU) for transient tachypnea of the newborn (TTN) or phototherapy
* status of mother-baby bonding and breastfeeding

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) II or III term pregnant women aged ≥18 years scheduled to undergo elective CS under spinal anesthesia between June 2021 and June 2023 in Gazi University

Exclusion Criteria:

Parturients younger than <18 years old with fetal compromise, ASA IV or V physical status and emergency cases, medical contraindication to regional anesthesia particularly spinal block

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — older than 18 years of age
Enrollment: 450 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
improved maternal recovery in term of ObsQoR in the ERAS pathway | From enrollment to the end of ERAS or control postpartum 24 hours
  Primary outcome measure is described as maternal recovery outcome measure determined by obstetric quality recovery score (ObsQoR) which has been known as a patient reported outcome mesaure (PROM) and neonatal outcome assessed by pediatricians.
  ObsQoR-11 scores with Likert scale corresponds to; zero being very poor and 110 being excellent

SECONDARY OUTCOMES:
implementation of maternal ERAS protocol improves newborn nutrition and breastfeeding | From enrollment to the end of ERAS or control postpartum 24 hours
  improved neonatal outcome in the ERAS pathway; nutrition-breastfeeding, higher number of newborns having full breast feeding than formula feeding

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine Department of Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be available when our work is published for 10 years .

REFERENCES:
- [Derived] Ozdemir MG, Gunaydin B, Bayram M, Hirfanoglu IM. Effect of enhanced recovery after surgery (ERAS) protocol on maternal and fetal outcomes following elective cesarean section: an observational trial. BMC Pregnancy Childbirth. 2025 Apr 29;25(1):517. doi: 10.1186/s12884-025-07583-3. PMID 40301800